CLINICAL TRIAL: NCT04376957
Title: Pilot Study of an Oral Chemotherapy Teaching Tool to Improve Adherence in Patients With Multiple Myeloma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hamilton Health Sciences Corporation (Other)
Responsible Party: Principal Investigator, Hira Mian, Hematologist, Juravinski Cancer Center Assistant Professor, Department of Oncology, McMaster University, Hamilton Health Sciences Corporation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 9495
Record Dates: First submitted 2020-04-26; First posted 2020-05-06 (Actual); Last update posted 2020-05-06 (Actual); Status verified 2020-05

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Intervention Model Description: Patients will be randomized to standard of care counselling done for oral myeloma medications or will be counselled using the novel teaching tool MASCC Oral agent Teaching Tool (MOATT). Standard of care consists of standard counselling and written materials provided by the oncologist or pharmacy (e.g. instructions and information on the regimen, common side effects, symptom management, medication safety and how to contact a clinician for any problems encountered).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Counselled with Current Standard Care (Active Comparator): Standard of care consists of standard counselling and written materials provided by the oncologist or pharmacy (e.g. instructions and information on the regimen, common side effects, symptom management, medication safety and how to contact a clinician for any problems encountered).
  Interventions: Behavioral: Standard of care consisting of standard counselling
- Counselled with MASCC Oral agent Teaching Tool (MOATT) (Experimental): This group will receive counselling using the MASCC Oral Agent Teaching Tool and be compared with the standard of care counselling.
  Interventions: Behavioral: Multinational Association of Supportive Care in Cancer Oral agent Teaching Tool

INTERVENTIONS:
Behavioral: Multinational Association of Supportive Care in Cancer Oral agent Teaching Tool — This tool was developed by an expert panel of oncology nurses and was further revised following external review of health care providers world-wide. This tools involves four key modules 1) patient's baseline knowledge, 2) patient education of oral cancer drugs 4) patient education tailored to a specific cancer drug 4) evaluation of the educational material.
  It was originally studied in 30 patients with lung cancer and was shown to be feasible with acceptable knowledge retention. Similarly, in a single center cohort study of general oncology patients, medication adherence self-efficacy appeared to improve with MOATT. The MOATT interventional tool incorporates key components of patient education and also has the advantage of being a potentially feasible tool that can be incorporated into future routine clinical practise.
  Other Names: MOATT
  Arms: Counselled with MASCC Oral agent Teaching Tool (MOATT)
Behavioral: Standard of care consisting of standard counselling — Consists of instructions and information on the regimen, common side effects, symptom management, medication safety and how to contact a clinician for any problems encountered.
  Arms: Counselled with Current Standard Care

SUMMARY:
Multiple Myeloma is an incurable cancer. Therapies for it include oral chemotherapy pills. It is unknown whether patients regularly and correctly take these anti-myeloma pills. This study wants to measure the rate of adults with MM taking anti-myeloma pills correctly. The investigators also want to use a teaching tool to see if it will help patients feel more satisfied and more confident in taking their anti-myeloma pills correctly. The investigators hope to use this data from this small study to eventually do a larger study in this area.

DETAILED DESCRIPTION:
The prevalence of patients with myeloma utilizing orally-administered myeloma therapy (OMT) is expected to continuously rise within Canada. The MASCC Oral agent Teaching Tool (MOATT) interventional tool relies on the concept of improved patient education in turn leading to improved adherence. Although the MOATT intervention is currently endorsed by Cancer Care Ontario, there is no data using the MOATT intervention in patients with myeloma or within Canada. Prior to embarking on a larger, multi-center study, a pilot study is necessary to 1) understand the feasibility, acceptability of the MOATT intervention and its preliminary efficacy 2) to determine the rates of adherence to OMT and explore factors associated with non-adherence and 3) to determine the feasibility of a larger multi-centre trial.

ELIGIBILITY:
Inclusion Criteria:

* Will include adults (age>18) with multiple myeloma who will be initiating OMT (lenalidomide or pomalidomide in the next 6 months) for either newly diagnosed, maintenance-phase or relapsed myeloma at the JCC

Exclusion Criteria:

* Patients who reside in a facility in which their medications are administered to them (such as a nursing home)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-08-01 (Estimated); Primary Completion 2022-02-01 (Estimated); Study Completion 2022-02-01 (Estimated)

PRIMARY OUTCOMES:
Personal Patient Preference Towards Using the MOATT Intervention assessed by a 5 point Likert scale. | 18 months from study recruitment date.
  Patient's preference and acceptability of using the MOATT intervention will be assessed using a 5 point Likert Scale after the intervention is completed. A higher score means a higher level of personal satisfaction and acceptance of the MOATT intervention.

SECONDARY OUTCOMES:
Objective adherence rate of medication assessed by number of cap openings. | 18 months from study recruitment date.
  All patients will be using the Medication Event Monitoring System (MEMS) pill cap and bottle which electronically records the date and time of the bottle opening to monitor adherence every month.
Self Reported Adherence Rate assessed by Brief Adherence Rating Scale (BARS). | 18 months from study recruitment date.
  Brief Adherence Rating Scale (BARS) is a self-reported administered medication adherence assessment. It consists of three questions and an overall visual analog rating scale that will be administered every month.
Toxicities of Oral Myeloma Treatment assessed by the Patient Reported Outcomes Common Terminology Criteria for Adverse Events (PRO-CTCAE tool). | 18 months from study recruitment date.
  PRO-CTCAE is a patient-reported outcome (PRO) measurement system developed to evaluate symptomatic toxicity in patients on cancer clinical trials. This will be administered every month.

CONTACTS AND LOCATIONS:
Overall Officials: Hira Mian, MD, Principal Investigator — Juravinski Cancer Center

IPD SHARING:
Plan to Share IPD: No